CLINICAL TRIAL: NCT00988195
Title: Recombinant Human Arginase I (rhArgI) for Patients With Advanced Hepatocellular Carcinoma (HCC): An Adaptive Design Dose Escalation Trial With Addition of Standard Doxorubicin Treatment
Brief Title: Study of Pegylated Human Recombinant Arginase for Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Cancer Treatment International Limited (Industry)
Collaborators: The University of Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKCTR-503; PR/CT205/07 (Other: Department of Health, HKSAR)
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Neoplasm; Hepatocellular Carcinoma
Keywords: Neoplasm; Hepatocellular Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular | interventions — BCT-100; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEG-BCT-100 (Experimental): Pegylated Recombinant Human Arginase I
  Interventions: Biological: Pegylated Recombinant Human Arginase I; Drug: Doxorubicin

INTERVENTIONS:
Biological: Pegylated Recombinant Human Arginase I — Week 1 (Single Dose); Weeks 3 - 11 (Weekly Dose x 8 weeks)in 8 escalation doses
  Other Names: PEG-BCT-100
Drug: Doxorubicin — Weeks 13-24 (once every 3 weeks)
  Other Names: Adriamycin

SUMMARY:
The purpose of this study is to determine whether recombinant human arginase (PEG-BCT-100) is safe and effective in the treatment of advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The primary objectives of this study are:

* To establish a safe dose level for weekly intravenous administration of PEG- BCT-100 (rhArgIpeg5000) based on clinical and laboratory safety assessments following a range of doses (from 500 to >5000 U/kg).
* To define the optimal biological dose (OBD) of PEG-BCT-100 based on the pharmacodynamics (PD) of arginine depletion (ADD) relative to plasma PK of PEG- BCT-100.
* To evaluate any objective tumor responses to PEG-BCT-100 in HCC patients receiving weekly doses of PEG-BCT-100 alone and in combination with standard doses of doxorubicin

Secondary objectives of this study are:

* To define any toxicities associated with the metabolic and cellular alterations of ADD relative to dose and PK of PEG-BCT-100 (rhArgIpeg5000).
* To develop a safe and biologically active dose and schedule for PEG-BCT-100 treatment in phase 2 trials, either as monotherapy or in combination with best standard of care chemotherapy.
* To confirm the safety and initial anti-tumor activity of the preferred dose and regimen of PEG-BCT-100 in 18 additional patients with advanced HCC

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HCC according to the European Association for the Study of the Liver criteria
* Known underlying HCC etiology specified by hepatitis B, hepatitis C, post alcoholic cirrhosis, or other
* HCC lesion(s) which are not resectable and which are measurable by C-T scan
* Progression of or non-response of HCC lesions after treatments which are considered best standard of care - surgical resection, radiofrequency ablation, chemoembolization
* No cancer treatment or surgery within the prior 4 weeks, either chemotherapy, targeted biologic or enzymes, either approved or investigational;
* Males or females from 18 to 75 years-old, inclusive;
* Ability and willingness to provide written informed consent;
* Karnofsky performance status of 80% or above and expected survival of more than 12 weeks; and,
* Negative urine pregnancy test, if female, and willingness to use an effective method of contraception during the entire study period

Exclusion Criteria:

* Advancing liver failure indicated by uncontrolled ascites, pleural effusions, encephalopathy, or a Child-Pugh score of C
* Significant hepatic, renal or bone marrow dysfunction indicated by total bilirubin >40 µmol/L, evidence of bile duct obstruction, serum albumin <30 g/L, serum SGOT >5 x upper limit of normal, ANC <1.0 x 10^9/L, platelets <100 x 10^9/L, or INR >2.0
* Significant cardiac or pulmonary disease defined by New York Heart Association (NYHA) Class III or IV, VEF <50% by echo or MUGA, or a history of myocardial infarction within the past 6 months, significant unstable arrhythmia or evidence of ischemia on ECG
* Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Significant active infection including HIV requiring oral or parenteral anti-infective therapies;
* Use of investigational drug(s) within 4 weeks of enrollment; or,
* Prior treatment with arginine depleting agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Plasma arginase and arginine levels,as well as tumour response, i.e. an effect on growth in the milieu of arginine depletion. | 24 weeks

SECONDARY OUTCOMES:
Overall Survival, Time to Progression | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie TP Poon, Prof, Principal Investigator — Division of Hepatobiliary and Pancreatic Surgery, Department of Surgery, The University of Hong Kong
Locations (1):
- Division of Hepatobiliary and Pancreatic Surgery, Department of Surgery, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- See also: HKCTR-503 — http://www.hkclinicaltrials.com/